CLINICAL TRIAL: NCT01950806
Title: The Effect of Pecans on Biomarkers of Risk for Cardiovascular Disease and Diabetes: A Controlled Feeding Trial in Overweight/Obese Adults With Central Adiposity
Brief Title: The Effect of Pecans on Biomarkers of Risk for Cardiovascular Disease and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Pecan Shellers Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB10998
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease Risk; Type 2 Diabetes Risk
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Pecan-containing diet (Active Comparator): Test diet containing 1.5 oz pecans/2000 kcal/day for 28 days
  Interventions: Other: Pecan-containing diet
- Nut-free diet (Placebo Comparator): Placebo diet containing no nuts or nut products, and identical in total fat and fiber as the test diet, for 28 days
  Interventions: Other: Nut-free diet

INTERVENTIONS:
Other: Pecan-containing diet
  Other Names: Isocaloric diet containing 1.5 oz pecans per 2000 kcal per day for 28 days
  Arms: Pecan-containing diet
Other: Nut-free diet
  Other Names: Isocaloric diet absent nuts and matched for total fat and fiber for 28 days.
  Arms: Nut-free diet

SUMMARY:
The objective of this randomized, controlled feeding study is to investigate the potential health benefits of a pecan-containing diet. The investigators hypothesize the chronic consumption of pecans will improve an array of biomarkers related to cardiovascular disease and type 2 diabetes risk, including indices of oxidative stress, antioxidant activity, inflammation, endothelial function, and insulin resistance when compared with a control diet that is absent nuts.

ELIGIBILITY:
Inclusion Criteria:

* Men & postmenopausal women, age 50 years and over
* BMI 25-35 kg/m2
* Waist/hip >0.8 for women and >0.9 for men
* Blood pressure between 120/80 and 159/99

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Individuals taking estrogen
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Regular use of any stomach acid-lowering medications, laxatives (including fiber supplements) or anti-diarrheal medications (prescription or over-the-counter [OTC])
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, unstable thyroid disease
* Autoimmune disease: including rheumatoid arthritis, gout, lupus, HIV
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 159 mmHg and/or diastolic blood pressure > 99 mmHg
* Regular use of oral or injectable steroids
* Gain or loss of > 10% of body weight within previous 3 months; unwillingness to maintain your weight
* Regular daily intake of ≥ 2 alcoholic drinks
* Vegetarians
* Current allergy to any kind of nut
* Dietary supplement use, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) homeopathic remedies, probiotics, or fish oil (including cod liver oil), for one month prior to study admission

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of oxidative stress compared with control diet | Baseline and 4 weeks
Change in biomarkers of inflammation compared with control diet | Baseline and 4 weeks.
Change in biomarkers of endothelial function compared with control diet | Baseline and 4 weeks.
Change in biomarkers of antioxidant activity compared with control diet | Baseline and 4 weeks
Change in biomarkers of insulin resistance compared with control diet | Baseline and 4 weeks

SECONDARY OUTCOMES:
Change in blood pressure compared with control diet | Baseline and 4 weeks
Change in plasma lipid profile compared with control diet | Baseline and 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States